CLINICAL TRIAL: NCT03921684
Title: Phase II Trial to Evaluate the Addition of Nivolumab to Neoadjuvant Chemoradiation With FOLFOX for Locally Advanced Rectal Cancer
Brief Title: Trial of Nivolumab With FOLFOX After Chemoradiation in Rectal Cancer Patients
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Baruch Brenner (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor-Investigator, Baruch Brenner, Head, Department of Oncology, Davidoff Cancer Center, Rabin Medical Center, Beilinson Hospital, Rabin Medical Center
Organization: Rabin Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA209-8M4
Record Dates: First submitted 2019-04-14; First posted 2019-04-19 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Rectal Cancer
Keywords: Nivolumab; Chemoradiation; mFOLFOX6; rectal cancer; Anti-PD-1 antibody
MeSH Terms: conditions — Rectal Neoplasms | interventions — Capecitabine; Radiotherapy; Nivolumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neoadjuvant Treatment (Experimental): All subjects will receive chemoradiation followed by chemotherapy and nivolumab as neoadjuvant treatment
  Interventions: Drug: Capecitabine; Radiation: Radiation therapy; Drug: mFOLFOX6; Drug: Nivolumab

INTERVENTIONS:
Drug: Capecitabine — Capecitabine 825 mg/m2 orally twice-daily, 5 days a week for a total of 28 days, given with radiation therapy
  Other Names: Xeloda
Radiation: Radiation therapy — 1.8 Gy/day, 5 days a week for a total of 28 days, given with Capecitabine
Drug: mFOLFOX6 — oxaliplatin 85 mg/m2, leucovorin 400 mg/m2 and fluorouracil 400 mg/m2 IV, fluorouracil 2400 mg/m2 IV (a 46 hrs CI), day 1 of each treatment cycle, every 2 weeks, given with nivolumab
Drug: Nivolumab — Nivolumab 240mg IV, day 1 of each treatment cycle, every two weeks, given with mFOLFOX6
  Other Names: Opdivo

SUMMARY:
This is a phase II, prospective, open label, one-center study for evaluation of the addition of nivolumab to the chemotherapy phase of the neoadjuvant treatment for locally advanced rectal cancer patients. Subjects must have received no prior treatment for rectal cancer (chemotherapy, radiotherapy or surgery) and no prior treatment with checkpoint inhibitors.

Eligible subjects will receive chemoradiation for a period of 5 weeks, 6 cycles of chemo-immunotherapy (mFOLFOX6 + nivolumab) for a period of 12 weeks, once every 2 weeks, and will undergo surgery after 4 weeks.

Patients with cCR will be offered the alternative strategy of WW. Post-study systemic treatment, up to 4 cycles of mFOLFOX6, will be left to the discretion of the treating physician. This will be started 4-8 weeks post-operatively, or immediately after the demonstration of cCR in patients determined to undergo WW.

ELIGIBILITY:
Inclusion Criteria:

* Signed written IRB approved informed consent
* Age ≥ 18 years
* ECOG PS 0-1
* Subjects with histologically confirmed primary (non-recurrent) locally advanced rectal adenocarcinoma
* Stage T3-4 N0 or TX N+ according to baseline rectal EUS and PET-CT
* Patients who are planned for neoadjuvant chemoradiation and are surgical candidates
* No prior chemotherapy, radiotherapy or surgery for rectal cancer
* No prior radiotherapy to the pelvis, for any reason
* Presence of adequate contraception in fertile patients
* Women of childbearing potential must have a negative serum or urine pregnancy test within 24 hours prior to the start of study drug
* Women must not be breastfeeding
* Ability to swallow tablets
* No previous (within the last 5 years) or concurrent malignancies, with the exception of adequately treated cone-biopsied in situ carcinoma of the cervix or basal cell carcinoma of the skin

Exclusion Criteria:

* Active autoimmune disease. [Subjects with type I diabetes mellitus, hypothyroidism only requiring hormone replacement, skin disorders (such as vitiligo, psoriasis, or alopecia) not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll]
* Prior treatment with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-CTLA-4 antibody, or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways
* Known history of positive test for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS)
* Pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2019-04-10 (Actual); Primary Completion 2024-10-28 (Actual); Study Completion 2029-10 (Estimated)

PRIMARY OUTCOMES:
pathological complete response (pCR) rate | Time from start of neoadjuvant treatment until surgical resection, assessed up to 24 months
  pCR is defined when no tumor is found on pathology review of the surgical specimen (TRG -0)
Incidence of Treatment-Emergent Adverse Events (Safety) | Time from screening until the end of study drug administration, assessed up to 24 months
  Treatment-emergent AEs will be graded according to NCI CTCAE v4.0, vital signs and clinical laboratory
modified pathological complete response | Time from start of neoadjuvant treatment until surgical resection in operated patients (pCR) and long-term (≥12 months) clinical complete response (cCR) in unoperated patients, assessed up to 24 months.
  We defined a novel primary endpoint, combining pathological complete response (pCR) rate among operated patients and long-term (≥12 months) clinical complete response (cCR) rate for those electing watchful waiting, into a composite endpoint of modified pCR (mpCR) rate.

SECONDARY OUTCOMES:
Disease Free Survival (DFS) | Time from the first day of treatment to the first event of: loco-regional failure, metastatic recurrence, the appearance of a secondary colorectal cancer or death from any cause, assessed up to 42 months
  DFS will be censored for patients who are alive and free of progression at the time of last follow-up. DFS rate will be estimated using the Kaplan-Meier method
Overall Survival (OS) | The time interval between the first day of treatment and the date of death of any cause, assessed up to 66 months
  Patients who are still alive when last traced will be censored at the date of last follow-up. OS rate will be estimated using the Kaplan-Meier method

CONTACTS AND LOCATIONS:
Overall Officials: Baruch Brenner, Prof, Principal Investigator — Rabin Medical Center
Locations (1):
- Rabin Medical Center, Beilinson Hospital, Petah Tikva, Israel